CLINICAL TRIAL: NCT07028073
Title: Avapritinib Combined With Standard Therapy for the Treatment of Newly Diagnosed KIT Mutation Acute Myeloid Leukemia With t(8;21)(q22;q22.1); Inv(16)(p13.1q22) or t(16;16)(p13.1;q22): a Prospective, Multi-center, Single-arm, Two-cohorts Study
Brief Title: A New Treatment of Newly Diagnosed KIT Mutation CBF-Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Prof., The First Affiliated Hospital of Soochow University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-AML03
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia With T(8;21)(Q22;Q22); Acute Myeloid Leukemia With T(16;16)(P13;Q22); KIT Gene Mutation; Avapritinib

STUDY DESIGN:
Intervention Model Description: Phase 1: Study treatment will start at level 1, and the therapeutic level will be escalated or descalated depending on the appearance of DLT. DLT will be monitored during cycle 1.
  Phase I will consist of two parallel dose escalation cohorts, with consecutive assignment to each group. For the dose escalation, we will use two parallel groups following a standard "3+3" design. Patients will be assigned sequentially to each group: Group A receives avapritinib with the IA regimen for fit patients, and Group B receives the VA regimen for those unfit.
  Phase II includes two treatment arm groups (IA-based RP2D vs. VA-based RP2D). Patients will be enrolled at diagnosis, within a maximum 28-day screening period, and will be assessed for eligibility for intensive therapy and therefore assigned to a treatment arm. All screening activities will be performed after the patient's informed consent form is signed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (FIT): Avapritinib Combined Intensive Chemotherapy in patients with newly diagnosed AML (Experimental)
  Interventions: Drug: Group A (FIT): Avapritinib + IA regimen
- Group B (UNFIT): Avapritinib Combined Venetoclax/Azacitidine in patients with newly diagnosed AML (Experimental)
  Interventions: Drug: Group B (UNFIT): Avapritinib + VA regimen

INTERVENTIONS:
Drug: Group A (FIT): Avapritinib + IA regimen — Cytarabine 100mg/m² days 1-7 Idarubicin 12mg/m² days 1-3 Avapritinib orally on days 8-21 (28-day cycle)
  Other Names: Group A (Intensive chemotherapy)
  Arms: Group A (FIT): Avapritinib Combined Intensive Chemotherapy in patients with newly diagnosed AML
Drug: Group B (UNFIT): Avapritinib + VA regimen — Venetoclax 100mg day 1, 200mg day 2, 400mg days 3-28 Azacitidine 75mg/m² days 1-7 Avapritinib orally on days 8-21 (28-day cycle)
  Other Names: Group B (Non-intensive chemotherapy)
  Arms: Group B (UNFIT): Avapritinib Combined Venetoclax/Azacitidine in patients with newly diagnosed AML

SUMMARY:
The goal of this clinical trial is to learn if avapritinib combined with standard induction therapy works to treat newly diagnosed adult acute myeloid leukemia (AML) patients with KIT mutations and t(8;21)(q22;q22.1); inv(16)(p13.1q22) or t(16;16)(p13.1;q22). It will also investigate the safety and tolerability of this combination therapy. The main questions it aims to answer are:

To determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of avapritinib combined with chemotherapy by Dose-limiting toxicity (DLT).

Does this combination therapy improve the rates of minimal residual disease (MRD) negativity and long-term survival outcomes?

DETAILED DESCRIPTION:
The prognosis of CBF-AML patients with KIT mutation remains relatively poor. CBF-AML is a heterogeneous disease in which many altered molecular pathways could contribute to the prognosis of the disease. Thus, curative approaches have been based on standard and high-dose cytarabine regimens using high-dose chemotherapy. However, the high rate of relapses in these patients should stimulate the development of new regimens. In recent years, there has been a series of new drugs under development that allow the design of combination therapies in this population. These drugs have an acceptable toxicity profile and are able to improve the CR rate in this population. In this way, the standard therapy and a small molecular targeted agent (Avapritinib) could produce a powerful antileukemic effect, preventing the adaptive escape mechanisms of leukemic cells. The investigators have designed a phase I-II trial based on the combination of a three-drug regimen (IA: standard-dose cytarabine + darubicin) or (VA: Azacitidine + Venetoclax) combined with avapritinib, which in this population could be well tolerated by a sequential type administration. The first objective is to achieve rapid control of the disease and the recommended dose for Phase II, using two different schemes, one based on IA and the other on VA, by dose escalation in Phase I of the trial. The second goal is to prevent relapse through a consolidation and maintenance schedule. Phase II will study the efficacy and safety of the recommended dose for Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, both genders
* Diagnosis of acute myeloid leukemia according to WHO 2022 criteria
* Treatment-naive patients (hydroxyurea or low-dose cytarabine <0.5g cumulative dose allowed)
* Bone marrow detection of KIT mutations with concurrent t(8;21)(q22;q22.1) or RUNX1::RUNX1T1 fusion gene; or inv(16)(p13.1q22) or t(16;16)(p13.1;q22) or CBFβ::MYH11 fusion gene
* Life expectancy >12 weeks Group A: ≥18 and <65 years with ECOG 0-1; Group B: ≥65 years or ≥18 and <65 years with comorbidities (ECOG ≥2, cardiac disease, creatinine clearance 30-50ml/min, or mild hepatic impairment)
* Adequate organ function: bilirubin ≤2×ULN, ALT/AST ≤3×ULN (≤5×ULN if leukemic infiltration), creatinine clearance ≥30ml/min, left ventricular ejection fraction >45%

Exclusion Criteria:

* Known hypersensitivity to KIT inhibitors, cytarabine, idarubicin, venetoclax, azacitidine or similar agents
* Concurrent use of other KIT inhibitors (dasatinib, sorafenib, gilteritinib, midostaurin)
* Intracranial hemorrhage on imaging or unresolved prior intracranial bleeding
* Active uncontrolled infection
* Significant organ dysfunction: myocardial infarction, chronic heart failure, decompensated liver dysfunction, renal failure
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Recommended phase 2 dose (RP2D) | Approximately 6 months after first patient first visit (FPFV)
  Recommended phase 2 dose (RP2D) of IA-based and VA-based combination with avapritinib schedules
Phase II: MRD (Measure residual disease) negativity rate | Aproximatey 2 years after FPFV
  MRD negativity rate - proportion of patients achieving ≥3-log reduction in RUNX1::RUNX1T1 or CBFβ::MYH11 fusion gene levels by qPCR between the 1st and 2nd consolidation courses.

SECONDARY OUTCOMES:
Overall survival (OS) | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  Overall survival will be defined as the number of days from the start of treatment to the date of death. Subjects that have not died will be censored at the last known date to be alive. To estimate 1, 2 and 3 years progression-free survival.
Composite complete remission rate (CRc) | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  Composite complete remission rate (CRc) after one cycle of induction therapy
Adverse Event | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  Safety profile: incidence of grade 3-4 clinical adverse events and laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China